CLINICAL TRIAL: NCT00418496
Title: A Phase I Study of Bolus High Dose Interleukin-2 With Sorafenib (BAY 43-9006) in Patients With Unresectable or Metastatic Clear Cell Renal Carcinoma (RCC) and Metastatic Melanoma
Brief Title: Interleukin-2 With Sorafenib (BAY 43-9006) for Unresectable or Metastatic Clear Cell Renal Carcinoma (RCC) and Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Bayer (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Paul Monk, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06006; NCI-2011-03199 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Renal Cancer; Melanoma
Keywords: Unresectable; Metastatic
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Neoplasm Metastasis | interventions — aldesleukin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aldekleukin Plus Dose Escalation Sorafenib (Experimental): Patients will be admitted to a dedicated nursing unit for HD aldesleukin administration. Patients will receive bolus aldesleukin at a dose of 600,000 IU/Kg every eight hours on days 1-5 with a goal of 10-12 doses.
  Interventions: Drug: Aldesleukin; Drug: Sorafenib

INTERVENTIONS:
Drug: Aldesleukin — 600,000 IU/kg every 8 hours on days 1-5 (week 1) to a maximum of 12 doses. Another cycle of HD aldesleukin will be started on day 15 (week 3).
  Other Names: Proleukin
Drug: Sorafenib — To be initiated at a dose of 200 mg orally. Once it is determined that no further HD aldesleukin therapy will be given, sorafenib may be given daily at the FDA approved dose of 400 mg twice daily until there is lack of clinical benefit or intolerable side effects develop.
  Other Names: Nexavar

SUMMARY:
The primary objective of this study will be to determine the toxicity and Maximum Tolerated Dose (MTD) of the combination of high dose aldesleukin and sorafenib in previously untreated patients with metastatic or unresectable clear cell renal carcinoma (RCC) and metastatic melanoma.

DETAILED DESCRIPTION:
Rationale: Previous research indicates that high dose aldesleukin produces tumor regression through upregulation of the patients' immune system. Research suggests that sorafenib directly targets tumors by inhibiting angiogenic activity with possibly some cytotoxicity. Angiogenic refers to the formation of new blood vessels that support tumor growth. Cytotoxicity is the measurement of a chemical's ability to damage or kill cancer cells. Researchers have hypothesized that the complementary ways aldesleukin and sorafenib work, and their non-overlapping toxicity profiles, may create a reasonable combination for the treatment of metastatic renal cell carcinoma and metastatic melanoma. The current Phase I study will evaluate toxicity in patients through assessing various dose levels of sorafenib in combination with aldesleukin.

Purpose: The primary objective is to determine the maximum tolerated dose and characterize the toxicity of high dose aldesleukin and sorafenib in patients with unresectable or metastatic clear cell renal carcinoma and metastatic melanoma. Secondary objectives include determining progression free survival in patients, evaluating in a preliminary manner response rates, and assessing other measurements in study participants.

Treatment: Study participants will be given bolus high dose aldesleukin and sorafenib. Aldesleukin will be provided through intravenous infusions on days 1 through 5. Each 5 day treatment is considered a cycle. The second cycle of aldesleukin will start on day 15. Two cycles are considered 1 course. All study participants will be given the same dose level of aldesleukin. No dose reductions will be permitted. Sorafenib will then be administered on day 29. Since this study will assess the maximum tolerated dose of sorafenib, some study participants will receive different amounts of this drug compared to others depending upon when each individual enrolls in the study. Each group of 3 to 6 study participants will receive a higher dose of sorafenib until the maximum tolerated dose is established. Imagining studies will be performed to determine response to treatment during week 12. If the patient has stable or responding disease, a second course will be administered on the same schedule. Patients without disease response will be given one additional course of aldesleukin past maximal response. When it is decided that no further aldesleukin will be provided to patients, sorafenib at the Food and Drug Administration approved dose may be continued until there is a lack of clinical benefit or intolerable side effects develop. Several tests and exams will be given throughout the study to closely monitor patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed evidence of metastatic/ unresectable clear cell renal carcinoma.
* Patients must have metastatic melanoma with no brain metastases.
* Patients must have measurable disease.
* No prior systemic treatment (One prior systemic treatment is allowed for metastatic melanoma patients. Excluded prior therapies include prior high dose aldesleukin, sorafenib and DTIC/TMZ.)
* Age ≥ 18 years or older

Exclusion Criteria:

* Patients who are undergoing or have undergone surgery S weeks.
* Patients who are pregnant (because of possible side effects on the fetus) Effective contraception will be discussed with each patient.
* Patients with uveal melanoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-11-08 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 1 year
  Determine the MTD for high dose (HD) aldesleukin and sorafenib in patients with metastatic or unresectable clear cell renal cell carcinoma and metastatic melanoma

SECONDARY OUTCOMES:
Determine the progression free survival. | Up to 12 weeks
Evaluate in a preliminary manner the response rate. | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Monk, M.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Monk P, Lam E, Mortazavi A, Kendra K, Lesinski GB, Mace TA, Geyer S, Carson WE 3rd, Tahiri S, Bhinder A, Clinton SK, Olencki T. A phase I study of high-dose interleukin-2 with sorafenib in patients with metastatic renal cell carcinoma and melanoma. J Immunother. 2014 Apr;37(3):180-6. doi: 10.1097/CJI.0000000000000023. PMID 24598448
- See also: Jamesline 1-800-293-5066 — http://cancer.osu.edu